CLINICAL TRIAL: NCT04784312
Title: A Phase Ia Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Immunogenicity of a Single Dose of MW14 Injection in Healthy Subjects
Brief Title: A Clinical Study in Health Subjects to Evaluate 9MW1411 Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9MW1411-2020-CP101
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2021-12

CONDITIONS: Staphylococcus Aureus Infection
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW1411 injection (Experimental)
  Interventions: Combination Product: 9MW1411 injection
- 9MW1411 injection placebo (Experimental)
  Interventions: Combination Product: 9MW1411 injection placebo

INTERVENTIONS:
Combination Product: 9MW1411 injection — 9MW1411 injection
  Arms: 9MW1411 injection
Combination Product: 9MW1411 injection placebo — 9MW1411 injection placebo
  Arms: 9MW1411 injection placebo

SUMMARY:
This is a Phase 1, first time in human study enrolling approximately 42 healthy adult subjects (18-45 yrs) from one study site. The purpose of this study is to evaluate the safety, tolerability and PK of MW14 in healthy adult volunteers administered as a single IV dose compared with placebo, across 5 cohorts. The 5 dose cohorts will enroll sequentially. Subjects will be followed for safety from the time of Informed Consent through 85 days post dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 45 years (including 18 and 45 years).
2. Weight≥50.0 kg for males, or weight≥45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 26.0 kg/m2 (including cut-off value).
3. The medical history, physical examination, clinical laboratory tests and other tests related study show no abnormalities, or abnormalities without clinical significance.
4. Subjects do not have a pregnancy plan, have no sperm and egg donation plans during the screening period and the next 6 months, and take effective contraceptive measures voluntarily.
5. Are willing to follow study procedures, signed informed consent voluntarily, and ensure that he/she will complete the study according to the program requirements.

Exclusion Criteria:

Prior or current medical conditions:

1. Health status: clinically significant histories of heart, liver, kidney, digestive tract, nervous system, respiratory system, blood and lymphatic system, immune system, mental, metabolic, and bone abnormalities.
2. Subjects who have a history of allergies to biological agents or any drug components; those who have a history of allergies and judged by the investigator to be ineligible for enrollment.
3. Those who undergone acute infection within 2 weeks prior to screening.
4. Those with abnormalities in pulmonary imaging examination prior to screening and judged to be clinically significant by the investigator.
5. Those who have undergone surgery within 3 months prior to screening, or who plan to undergo surgery during the study.
6. Those who cannot tolerate venipuncture or have a history of needle-sickness and blood-sickness.
7. Those who have a history of drug abuse within 6 months prior to screening.
8. Use of illicit drugs within 3 months prior to screening.
9. Those who donated blood within 3 months prior to screening (including component blood), or massive blood loss (≥ 200 mL), or blood transfusions or use of blood products.
10. Subject (female) who is pregnant or lactating at screening or during the trial.
11. Subjects have a fertility plan or sperm or egg donation plan at screening and within the next 6 months.
12. Use of any prescription, over-the-counter, or Chinese herbal medicines within 2 weeks prior to screening.
13. Those who have been vaccinated within 4 weeks prior to screening or who are scheduled to be vaccinated during the study.
14. Those who have smoked more than 5 cigarettes per day within 3 months prior to screening.
15. Those who have consumed more than 14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 3 months prior to screening, or who cannot abstain from alcohol during the trial.
16. Those who have special dietary requirements and cannot accept a standard diet.
17. Those who have participated in drug or medical devices clinical trials within 3 months prior to screening.
18. Those who have previously used immunosuppressants or monoclonal antibodies for any reason.
19. Those with abnormal vital signs with clinical significance: diastolic blood pressure≤50 mmHg or ≥90 mmHg, pulse≤50 beats/min or ≥100 beats/min, body temperature (ear temperature) <35.5°C or >37.5°C, respiration>20 breaths/min. The specific situation will be comprehensively determined by the investigator.
20. Those with abnormalities in laboratory tests and auxiliary examinations that are judged by the investigator to be clinically significant.
21. Those who have one or more clinically significant tests of hepatitis B virological markers, hepatitis C virus antibodies, anti-human immunodeficiency virus antibodies, or anti-Treponema pallidum-specific antibodies.
22. Female subjects with a positive blood pregnancy test at screening.
23. Alcohol breath test results greater than 0.0 mg/100 ml or positive drug screening (morphine, icenarcotics [methamphetamine], ketamine, ecstasy [methylenedioxyamphetamine], cannabis [tetrahydrocannabinolate], erythroxylin).
24. Subjects who is inappropriate to participate in the trial due to any reasons as determined by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 12 weeks
  safety evaluation
Serious Adverse Event | 12 weeks
  safety evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China